CLINICAL TRIAL: NCT05061147
Title: A Single-arm, Multi-Center, Phase Ib/Ⅱ Clinical Trial of Max-40279-01 in Combination With Azacitidine (AZA) in Adult Patients With Myelodysplastic Syndrome (MDS) or Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
Brief Title: A Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Max-40279-01 in Combination With Azacitidine (AZA) in Patients With Myelodysplastic Syndrome (MDS) or Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-004
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Leukemia; Acute Myeloid Leukemia; Relapsed/Refractory Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Relapsed/Refractory Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Max-40279-01 in combination with Azacitidine (AZA) (Experimental): This is an open-label Phase Ib/II clinical study. The study will be conducted in two parts:
  Part I: Phase Ib dose escalation. Participants receive Max-40279-01 in combination with azacytidine (AZA), with different dose schedules.
  Part II: Phase II dose expansion. Participants divide into positive group and negative group according to whether FLT3 gene mutation occurs, approximately 40 people per group.
  All participants receive the recommended dose for Part 2 of Max-40279-01 with azacytidine (AZA).
  Interventions: Drug: MAX-40279-01

INTERVENTIONS:
Drug: MAX-40279-01 — Drug: AZA AZA will be administered at 75 mg/m^2 by subcutaneous injection for 7 consecutive days from D1 to D7 in 28-day treatment cycles.
  Other Name: Azacitidine
  Drug: Max-40279-01 Max-40279-01 will be administered as a combination of multiple oral capsules containing 5 and 25 mg. An alternate combination of 35 mg, 50 mg and 60 mg Max-40279-01 twice a day may be utilized.
  Other Name: NA
  Other Names: Azacitidine (AZA)

SUMMARY:
This study is a phase Ib/II study of Max-40279-01 in combination with Azacitidine (AZA) in patients with Myelodysplastic Syndrome (MDS) or Relapsed/Refractory Acute Myeloid Leukemia (R/R AML). This study include Phase Ib and Phase II study. The phase Ib study is designed to evaluate the safety and tolerability of MAX-40279-01 in combination with Azacitidine (AZA) in patients with Relapsed or Refractory AML. The phase II study is designed to preliminarily assess the efficacy and safety of Max-40279-01 in combination with Azacitidine (AZA) in patients with Myelodysplastic Syndrome (MDS) or Relapsed/Refractory Acute Myeloid Leukemia (R/R AML).

DETAILED DESCRIPTION:
This is a two-part study comprised of a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. A diagnosis of AML according to the World Health Organization (WHO) 2016 criteria with relapsed or refractory disease and have exhausted, or are ineligible for therapeutic options, or int-risk or high-risk or very high-risk MDS according to revised International Prognostic Scoring System (IPSS-R);
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Expected survival >3 months.
5. No radiotherapy, surgery or hormonal therapy for any kind of within 2 weeks prior to participating in this study. Patients must have fully recovered from the acute toxicities of any prior treatment with any anti-cancer drugs (including hypomethylating agents in MDS patients), radiotherapy or other anti-cancer modalities (i.e., returned to baseline status as noted before most recent treatment) for any tumors. Patients with persisting, stable chronic toxicities from such prior treatment ≤Grade 1 are eligible, but must be documented as such.
6. Signed informed consent form.

Exclusion Criteria:

1. Acute promyelocytic leukemia according to World Health Organization 2016 criteria
2. Known central nervous system involvement
3. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product
4. Known allergies, hypersensitivity, or intolerance to Max-40279-01 or AZA or the excipients of these treatments
5. Previously treated malignancies other than the current disease, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years at the trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Through study Part 1 completion, an average of 6 months
  To explore the maximum tolerable dose (MTD) of Max-40279-01 in combination with Azacitidine (AZA) for patients with r/r AML or MDS, the recommended phase II dose (RP2D).
Phase II dose (RP2D) | Through study Part 1 completion, an average of 6 months
  Recommended phase II dose (RP2D)
Overall survival(OS) | Up to 24 months
Rate of complete remission (CRc) | Up to 24 months
  including Complete Remission with incomplete Platelet recovery (CRp) and Complete Remission with incomplete hematologic recovery (CRi)

SECONDARY OUTCOMES:
Tmax | Approximately 4 weeks
  Time to maximum plasma concentration
Cmax | Approximately 4 weeks
  Maximum plasma drug concentration
AUC | Approximately 4 weeks
  Area under the time-concentration curve
t1/2 | Approximately 4 weeks
  Observed terminal half-life
Objective response rate (ORR) | 1 months (anticipated)
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on IRWG.
Safety and tolerability assessed by incidence and severity of adverse events | 24 months
  All grade ≥ 3 toxicities according to CTCAE (Common Terminology Criteria for Adverse Events) version 5 will be tabulated

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No